CLINICAL TRIAL: NCT04760717
Title: Regulating Blood Pressure During Recovery From Intracerebral Hemorrhage and Ischemic Stroke
Acronym: REDUCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000029811
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Intracerebral Hemorrhage; Ischemic Stroke; Spironolactone
MeSH Terms: conditions — Cerebral Hemorrhage; Ischemic Stroke | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spironolactone (Experimental): Participants randomized to the Spironolactone arm will be receiving Spironolactone in addition to their normal routine blood pressure treatment.
  Interventions: Drug: Spironolactone Pill
- Standard Care (No Intervention): Participants randomized to the Standard care arm will be receiving their normal routine blood pressure treatment.

INTERVENTIONS:
Drug: Spironolactone Pill — Participants randomized to the Spironolactone arm will be receiving Spironolactone in addition to their normal routine blood pressure treatment.
  Arms: Spironolactone

SUMMARY:
The purpose of this research study is to determine whether blood pressure treatment regimens with spironolactone are better than blood pressure treatment regimens without spironolactone at lowering blood pressure in stroke survivors.

DETAILED DESCRIPTION:
This is a pragmatic, randomized, open-label, blinded-endpoint trial comparing spironolactone-containing antihypertensive regimens versus standard antihypertensive regimens based on the 2017 AHA/ACC guidelines in stroke survivors.

This study will randomize a total of 200 patients, 100 white and 100 non-white patients, at least three weeks after last known normal or symptom discovery/onset of their stroke to an antihypertensive regimen with spironolactone once daily or standard BP control based on the 2017 AHA/ACC guidelines for 1 year.

Participants will undergo baseline testing for neurohormonal levels and will be followed for 12 months with regular assessment of home BP readings. The primary outcome of home systolic BP will be measured at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Symptomatic ICH confirmed by head CT or brain MRI during hospitalization OR ischemic stroke patients. Ischemic stroke will be defined by focal signs/symptoms of any duration associated with evidence of acute arterial infarction on neuroimaging or clinical evidence of cerebral focal arterial ischemic injury with symptoms persisting ≥ 24 hours.
3. Written, informed consent by patient or surrogate
4. Ability to comply with all study procedures and available for the duration of the study

Exclusion Criteria:

1. Secondary ICH due to trauma, vascular malformation, or tumor
2. Life expectancy < 1 year
3. eGFR <45
4. Serum potassium greater than or equal to the upper limit of normal of the lab on the two most recent consecutive potassium levels prior to enrollment
5. Known hypersensitivity to spironolactone
6. Upper arm greater than 17 inches in circumference
7. Pregnancy, planned pregnancy, or breastfeeding
8. Contraindication to discontinuing mineralocorticoid antagonist therapy for 3-12 months per the investigator's discretion (e.g., refractory proteinuria)
9. Systolic BP >200 mmHg or diastolic BP >110 mmHg at the time of randomization
10. Systolic BP <120 mmHg at the time of randomization
11. Any condition which, in the judgement of the investigator, increases the risk to the patient
12. History of Addison's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Average change in home systolic blood pressure at 3 months | Baseline, 3 month
  The average home systolic blood pressure will be measured using a home blood pressure cuff

SECONDARY OUTCOMES:
Proportion of patients achieving BP < 130/80 mm Hg | 3 months
  The proportion of patients achieving BP < 130/80 mm Hg at 3 months will be measured
Number of antihypertensive medications at 3 months | 3 months
  The number of antihypertensive medications at 3 months will be collected
Number of antihypertensive medications at 1 year | 1 year
  The number of antihypertensive medications at 1 year will be collected
Stroke, myocardial infarction, or death | 1 year
  Incidence of stroke of any type (ischemic or hemorrhagic), myocardial infarction, or death from any cause
Change in modified Rankin Scale score | Baseline, 1 year
  Measure of neurologic disability (0=no disability to 6=dead)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes